CLINICAL TRIAL: NCT01962701
Title: Fetal Copeptin After Oxytocin Challenge Test
Acronym: CopOCT
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: CopOCT
Record Dates: First submitted 2013-10-10; First posted 2013-10-14 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Pregnancy
Keywords: C-section

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — EDTA plasma of arterial umbilical cord blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- OCT-group: OCT prior to C-section
- None-OCT-group: No OCT prior to C-section

SUMMARY:
The relationship of uterine contractions on fetal copeptin levels in umbilical cord blood is studied.

DETAILED DESCRIPTION:
Background: Vaginal delivery evokes a dramatic surge in stress hormones facilitating the transition of the infant to extra-uterine life. Infants born by elective cesarean section (C-section) are known to have a higher risk for compromised birth adaptation. Labor is vital for vaginal delivery and triggers fetal stress hormone release. Fetal plasma copeptin, a surrogate marker of arginine vasopressin, has been found to be 100 to 1000-fold increased after vaginal delivery as compared to elective C-section. However, the relationship of labor intensity and fetal stress hormone release is largely unknown.

Objective: The purpose of this study is to determine fetal copeptin in newborns delivered by C-section to mothers who had an oxytocin challenge test (OCT) just prior to birth as compared to those without OCT.

Protocol: Pregnant women at term are eligible to participate if no uterine contractions are reported within the last 24 hours and no contractions are recorded in cardiotocogram over 30 minutes. Further inclusion and exclusion criteria see below. After written informed consent, all participants get an infusion line and participants receive OCT or placebo. The OCT is standardized as follows: 5 IE Syntocinon (oxytocin) in 500 mL Ringer, infusion rate begins with 12 ml/h and is increased by steps of additional 12 ml/h until three contractions within ten minutes are recorded. Subsequently, infusion is stopped. The placebo is Ringer infusion without Syntocinon. C-section is done about 1 to 3 hours after OCT or placebo and arterial umbilical cord blood is collected at birth. Maternal and newborn data are recorded within the first few days after birth, including maternal blood loss, neonatal adaptation, and postnatal weight loss.

ELIGIBILITY:
Inclusion criteria:

* Singleton pregnancy
* Gestational age more than 36 weeks
* No contractions reported within the last 24 hours
* No contractions recorded by 30 min cardiotocogram prior to oxytocin challenge test

Exclusion criteria:

* All contraindications for labor, including placenta praevia
* Serious fetal malformations
* Anhydramnios
* Oligohydramnios
* IUGR < 5. percentile
* Presence of any contractions
* Suspicious or pathological fetal heart rate tracing (cardiotocogram)
* Any clinical or biochemical signs of maternal infection
* Breech presentation
* More than 1 C-section in history

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Primary care hospital, healthy pregnant women presenting for delivery at term
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2013-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Fetal plasma copeptin concentration | 30 min after delivery
  To be determined in arterial umbilical cord blood at birth

CONTACTS AND LOCATIONS:
Overall Officials: Tilo Burkhardt, MD, Principal Investigator — University Hospital Zurich, Department of Obstetrics
Locations (1):
- University Hospital Zurich, Department of Obstetrics, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wellmann S, Koslowski A, Spanaus K, Zimmermann R, Burkhardt T. Fetal Release of Copeptin in Response to Maternal Oxytocin Administration: A Randomized Controlled Trial. Obstet Gynecol. 2016 Oct;128(4):699-703. doi: 10.1097/AOG.0000000000001594. PMID 27607861